CLINICAL TRIAL: NCT02791828
Title: Creation and Validation of an Instrument for Measuring the Quality of Experience of a Hemodialysis of Chronic Renal Insufficiency Subject
Brief Title: Creation and Validation of a Questionnaire to Measure the Feelings of a Chronic Renal Insufficiency Person During His Hemodialysis
Acronym: VecuHD
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: CHU de Reims (Other)
Responsible Party: Sponsor
Other Study IDs: PR16030
Record Dates: First submitted 2016-05-27; First posted 2016-06-07 (Estimated); Last update posted 2016-06-07 (Estimated); Status verified 2016-05

CONDITIONS: Chronic Renal Insufficiency
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
Chronic Hemodialysis is a treatment for kidney failure. It involves the construction of three treatment sessions per week extrarenal lasting 4 hours each. This treatment is necessary but it has an impact on the quality of life of patients.The investigators believe that to improve the overall quality of life in hemodialysis patients, the quality of each hemodialysis session must be improved. The quality criterion is not only medical, it must also take into account the patient's perception about the course of its meeting : that's what we call quality of experience of the dialysis session. Our daily healthcare practice shows that each hemodialysis session is experienced differently by the patient according to different factors : physical, psychological, relational, technical, temporal. The quality of the experience of a hemodialysis session could be positively influenced by the use of supplements occupational assets or liabilities, for improving patient satisfaction or by enhancing its relationship with the staff. Indeed, a preliminary study ( in the nephrology unit of our establishment in January 2012) of 8 patients undergoing active occupational educational activity during hemodialysis, showed that the experience of the hemodialysis session was potentially improvable (experienced patients improved, reduced cramps ... ). However, to assess the impact of such measures on the lives of the dialysis session and the quality of life in general, the investigators need to measure the quality of living of a dialysis session. There is not, at present, specific tool to measure the quality of the experience of a hemodialysis session. This tool would measure the impact of a caregiver support occupational during dialysis sessions. The main objective of this study is to create and validate an instrument to measure the quality of living of a hemodialysis of chronic renal insufficiency subject.

DETAILED DESCRIPTION:
Chronic Hemodialysis is a treatment for kidney failure. It involves the construction of three treatment sessions per week extrarenal lasting 4 hours each. This treatment is necessary but it has an impact on the quality of life of patients. Indeed , the 2005 "REIN quality of life" report demonstrates that quality of life of people with kidney failure is impaired, especially in physical and general component. The investigators believe that to improve the overall quality of life in hemodialysis patients, we must improve the quality of each hemodialysis session. The quality criterion is not only medical, it must also take into account the patient's perception about the course of its meeting : that's what we call quality of experience of the dialysis session. Our daily healthcare practice shows that each hemodialysis session is experienced differently by the patient according to different factors : physical, psychological, relational, technical, temporal. The quality of the experience of a hemodialysis session could be positively influenced by the use of supplements occupational assets or liabilities, for improving patient satisfaction or by enhancing its relationship with the staff. Indeed, a preliminary study ( in the nephrology unit of our establishment in January 2012) of 8 patients undergoing active occupational educational activity during hemodialysis, showed that the experience of the hemodialysis session was potentially improvable (experienced patients improved, reduced cramps ... ). However, to assess the impact of such measures on the lives of the dialysis session and the quality of life in general, we need to measure the quality of living of a dialysis session. There is not, at present, specific tool to measure the quality of the experience of a hemodialysis session. This tool would measure the impact of a caregiver support occupational during dialysis sessions. Objectives: The main objective of this study is to create and validate an instrument to measure the quality of living of a hemodialysis of chronic renal insufficiency subject. This will be done in 3 steps, 1st step in establishing an item bank , second stage of construction and final calibration tool, and third step of psychometric validation of the questionnaire. Material and Methods : To date, no measure of the quality of living of a hemodialysis session is available and validated. The investigators intend to build and validate a quality instrument experienced a hemodialysis session for people with chronic kidney failure. The study will be conducted in three stages: - First step: the development of a bank of issue items qualitative research on the subject ( literature review , expert opinion ) and direct collection by focus group with people with CKD . - Second step: operationalization of the measuring tool (reduction of item bank , grouping of items ) with validation of the pre- final tool by individual statistical techniques (content validity , perceived validity, structure validity, internal consistency) .- Third stage: the psychometric validation of the final tool will be made after a survey conducted on subjects with CKD , aged 18 and older . These patients will be enrolled in the hemodialysis centers participants during a usual hemodialysis session. A total of 30 patients will be interviewed for the qualitative step of developing a bank of items and then again 30 patients will participate in the validation of the pre-final tool. Then 100 patients will be included to develop the final measurement tool and structure validation and 150 patients will be asked to analyze the psychometric properties (validity, reliability and sensitivity to change).The last two stages of this work will multicentric. For the development of the item bank and meter validation of the final tool of cross-sectional surveys are sufficient. For the validation phase , a longitudinal follow-up will be required , with a collection on day 0 , 7 day intervals (test - retest) and a collection to 6 months for the predictive validity of the assessment phase and sensitivity change. Analysis of the results will help define the applicability criteria and acceptability to know the validity of the specific instrument that is to say, its content validity, perceived validity, structure validity, discriminant validity, reliability explored by internal consistency and stability over time. Longitudinal follow-up of patients is expected to also assess the predictive validity and sensitivity to change. Statistical analysis plan: Statistical analysis of the data will use the so-called classical methods adapted. The study of the applicability of the instrument involves the description of relevant parameters. The validity of the instrument will use the following techniques: statistical techniques implement the factor analysis for the reduction of the items, check the dimensionality of fields, and check the structural validity. Analysis of variance or its equivalent for the study of discriminative ability. Reliability will be explored by the Cronbach alpha for internal consistency. For the study of reproducibility, the intraclass correlation coefficient is used. Multivariate analysis by Cox model or logistic regression will be performed to investigate the predictive validity and sensitivity to change. Expected results and prospects : The investigators believe that improving each hemodialysis session individually could ultimately improve the overall quality of life of patients. Hemodialysis treatment is palliative treatment (curative treatment is kidney transplantation), the medical teams have only as care option, improving the quality of sessions and therefore the experience of dialysis sessions. The investigators believe that the creation of a measurement tool and its validation are essential for the future evaluation of our actions. This tool will be useful for the entire Francophone community nephrologist .

ELIGIBILITY:
Inclusion Criteria:

Will be included in the study , patients :

* From 18 years or more;
* Achieved with chronic renal failure;
* Under hemodialysis;
* fluent in French .
* With a social security scheme.

Will not be included in the study , patients :

* Having cognitive problems hindering understanding of the tool.
* Having participated in Phase I of the research project.
* Under Backup Justice (guardianship)."

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients will be recruited volunteers hemodialysis centers
Sampling Method: Non-Probability Sample
Enrollment: 320
Dates: Start 2016-03; Primary Completion 2019-01 (Estimated); Study Completion 2019-07 (Estimated)

PRIMARY OUTCOMES:
quality of life of a hemodialysis of chronic renal insufficiency subject | 3 years

CONTACTS AND LOCATIONS:
Locations (1):
- Chu Reims, Reims, France